CLINICAL TRIAL: NCT01787760
Title: Controlling Myopia Progression With Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-1561AC
Record Dates: First submitted 2013-02-06; First posted 2013-02-11 (Estimated); Results first posted 2015-07-29 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Test Soft Contact Lens B (Experimental): Lenses will be worn in a daily disposable modality
  Interventions: Device: Test Soft Contact Lens B
- Test Soft Contact Lens C (Experimental): Lenses will be worn in a daily disposable modality
  Interventions: Device: Test Soft Contact Lens C
- Spectacle Lenses (Active Comparator): Control spectacle lenses worn daily.
  Interventions: Device: Active Comparator

INTERVENTIONS:
Device: Test Soft Contact Lens B — Test lenses to be worn in daily wear modality
  Arms: Test Soft Contact Lens B
Device: Test Soft Contact Lens C — Test lenses to be worn in a daily wear modality
  Arms: Test Soft Contact Lens C
Device: Active Comparator — Control spectacle lenses to be worn in a daily wear modality
  Arms: Spectacle Lenses

SUMMARY:
This study is to investigate whether novel soft contact lens optical designs can slow myopia progression.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be between 8 and 12 years of age and of Asia origin.
2. The subject's best sphere contact lens correction must lie between -0.75D (best of the two eyes) and -5.00D (worst of the two eyes)
3. Astigmatism must be less than or equal to 1.00D
4. Less than 1.00D difference in spherical equivalent between the two eyes
5. The subject must have a best-corrected visual acuity of 20/25 and spherical equivalent refraction visual acuity of 20/25 or better in both eyes
6. The subject must have at least 8D of accommodation.
7. The subject's parent or legal guardian must read and sign the STATEMENT OF INFORMED CONSENT and the subject must read and sign the Child's Assent Form and be provided a copy of each form
8. The subject must appear able and willing to adhere to the instructions set forth in the clinical protocol

Exclusion Criteria:

1. Ocular or systemic allergies or diseases that may interfere with contact lens wear
2. Systemic disease or autoimmune disease or use of medication (e.g. antihistamines), which may interfere with contact lens wear.
3. Clinically significant (grade 3 or 4) tarsal abnormalities or bulbar injection that might interfere with contact lens wear.
4. Clinically significant (grade 3 or 4) corneal edema, corneal vascularization, corneal staining, or any other abnormality of the cornea, which may contraindicate contact lens wear.
5. Any ocular infection.
6. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
7. Any infectious disease (e.g. hepatitis, tuberculosis) or immunosuppressive disease (e.g. HIV).
8. Diabetes.
9. Anismetropia.
10. Astigmatism of greater than 1.00D in either eye.
11. Eye injury or eye surgery within eight weeks immediately prior to enrollment for this study.
12. Previous refractive surgery, rigid contact lens wear, orthokeratology, keratoconus, or other corneal irregularity in either eye
13. Strabismus in either eye
14. Pupil or lid abnormality or infection in either eye
15. Central corneal scar and aphakia in either eye
16. Contraindications to contact lens wear such as dry eye or history of prior unsuccessful contact lens wear
17. History of participation in clinical trials aimed to control myopia progression
18. Surgically altered eyes, ocular infection of any type, ocular inflammation
19. Subject has anterior chamber angle grade 2 or narrower

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 221 (Actual)
Dates: Start 2007-04-01 (Actual); Primary Completion 2010-04-01 (Actual); Study Completion 2010-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Kowloon, Hong Kong

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of those 221 screened subjects, 56 were ineligible to participate in the study and 13 were eligible but not randomized to the study lens groups.
Period: Overall Study
Arm/Group | Test Soft Contact Lens B | Test Soft Contact Lens C | Spectacle Lenses
Started | 51 | 50 | 51
Completed | 25 | 34 | 46
Not Completed | 26 | 16 | 5
Not completed — Anisometropia > -1.00D in spherical equi | 1 | 0 | 0
Not completed — Decompensated on left exotropia | 0 | 0 | 1
Not completed — Dryness | 0 | 1 | 0
Not completed — Relocation | 1 | 1 | 0
Not completed — Lens discomfort | 3 | 0 | 0
Not completed — Lens handling difficulty | 1 | 2 | 0
Not completed — Protocol Violation | 6 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 1 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Stroke | 1 | 0 | 0
Not completed — Unsatisfactory lens fitting performance | 3 | 6 | 0
Not completed — Unsatisfactory physiological response | 2 | 4 | 0
Not completed — Unsatisfactory visual response | 1 | 1 | 0
Not completed — Near vision blur | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline summary was conducted on all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Soft Contact Lens B | Test Soft Contact Lens C | Spectacle Lenses | Total
Number analyzed (Participants) | 51 | 50 | 51 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 51 | 50 | 51 | 152
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.5 (1.1) | 9.6 (1.1) | 9.5 (1.1) | 9.5 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 31 | 23 | 72
  Male | 33 | 19 | 28 | 80
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Hong Kong | 51 | 50 | 51 | 152

OUTCOME MEASURES:

1. Primary Outcome: Axial Length (Axial Elongation)
Description: Axial Length was measured with the IOLMaster at baseline, and then every 6 months throughout the course of the study. Five measurements were collected for each eye at each visit and the average of the 5 measurements were used for the analysis. Higher values of axial elongation indicate worse vision.
Time Frame: Baseline and every 6 months post-baseline up to 3 years
Population: Analysis was conducted on all randomized subjects who have at least one data point.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Units Other Than Participants: eyes
Arm/Group | Spectacle Lenses | Test Soft Contact Lens B | Test Soft Contact Lens C
Number analyzed (Participants) | 48 | 36 | 37
Number analyzed (eyes) | 96 | 70 | 74
millimeter (mm)
  Change from baseline 6 months: number analyzed (eyes) | 96 | 70 | 72
  Change from baseline 6 months | 0.158 (0.0981) | 0.144 (0.0834) | 0.121 (0.0749)
  Change from baseline 12 months | 0.242 (0.1448) | 0.236 (0.1267) | 0.222 (0.1288)
  Change from baseline 18 months; N=92, N=54, N=72: number analyzed (eyes) | 92 | 54 | 72
  Change from baseline 18 months; N=92, N=54, N=72 | 0.348 (0.2129) | 0.355 (0.1837) | 0.344 (0.1676)
  Change from baseline 24 months; N=92, N=54, N=72: number analyzed (eyes) | 92 | 54 | 72
  Change from baseline 24 months; N=92, N=54, N=72 | 0.455 (0.2520) | 0.409 (0.2247) | 0.445 (0.2444)
  Change from baseline 30 months: number analyzed (eyes) | 70 | 40 | 58
  Change from baseline 30 months | 0.565 (0.2941) | 0.512 (0.2634) | 0.511 (0.2564)
  Change from baseline 36 months: number analyzed (eyes) | 16 | 8 | 10
  Change from baseline 36 months | 0.640 (0.3199) | 0.634 (0.3249) | 0.512 (0.3072)

2. Primary Outcome: Spherical Equivalent Refraction
Description: Spherical Equivalent Refraction was computed from the sphero-cylindrical refraction measured with an open-field auto refractor. The median of 3 repeated measurements, each of which was the average of 3 consecutive readings, was used for the analysis. Higher values of spherical refraction indicate progression in Myopia.
Time Frame: Baseline and every 6 months post-baseline up to 3 years
Population: Analysis was conducted on all randomized subjects who have at least one data point.
Measure: Mean (Standard Deviation); unit: diopter (D)
Units Other Than Participants: eyes
Arm/Group | Spectacle Lenses | Test Soft Contact Lens B | Test Soft Contact Lens C
Number analyzed (Participants) | 48 | 36 | 37
Number analyzed (eyes) | 96 | 70 | 72
diopter (D)
  Change from baseline 6 months: number analyzed (eyes) | 96 | 70 | 70
  Change from baseline 6 months | -0.238 (0.3443) | -0.327 (0.3038) | -0.230 (0.3436)
  Change from baseline 12 months: number analyzed (eyes) | 96 | 68 | 72
  Change from baseline 12 months | -0.417 (0.4557) | -0.456 (0.3733) | -0.429 (0.4199)
  Change from baseline 18 months: number analyzed (eyes) | 92 | 54 | 70
  Change from baseline 18 months | -0.562 (0.5841) | -0.692 (0.3965) | -0.720 (0.4988)
  Change from baseline 24 months: number analyzed (eyes) | 92 | 54 | 70
  Change from baseline 24 months | -0.776 (0.6185) | -0.781 (0.4447) | -0.861 (0.5504)
  Change from baseline 30 months: number analyzed (eyes) | 70 | 40 | 56
  Change from baseline 30 months | -0.966 (0.7592) | -1.000 (0.5485) | -1.003 (0.6829)
  Change from baseline 36 months: number analyzed (eyes) | 16 | 8 | 10
  Change from baseline 36 months | -1.073 (0.9922) | -1.266 (0.3193) | -0.824 (0.8244)

ADVERSE EVENTS:
Groups:
- Not Randomized: Subjects who met the all study eligible criteria but did not randomize to the study arm.
Arm/Group | Spectacle Lenses | Test Soft Contact Lens B | Test Soft Contact Lens C | Not Randomized
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51 | 0/50 | 0/13
Other Adverse Events (participants affected / at risk) | 0/51 | 7/51 | 4/50 | 0/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spectacle Lenses (N=51) | Test Soft Contact Lens B (N=51) | Test Soft Contact Lens C (N=50) | Not Randomized (N=13)
Slit-lamp finding (Eye disorders) | 0 (0) | 7 (10) | 4 (5) | 0 (0) — Slit Lamp findings Grade 2 or less requiring treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes